CLINICAL TRIAL: NCT01764438
Title: The Incidence of Change in BCLC Stage by add-on Primovist-enhanced MRI During Initial Staging Work-up in HCC Patients Who Can be Candidates for Curative Treatment by Liver Dynamic CT: A Prospective Multicenter Study
Brief Title: Utility Study of Primovist-MRI on HCC Staging
Acronym: PrimovistMRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INBU study; INBU study group (Registry Identifier: INBU group for the study of the liver)
Record Dates: First submitted 2013-01-01; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2012-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- very early or early staged patients: Performance of Primovist-enhanced MRI in HCC patients with very early or early stage disease, but with no suspicious HCC by liver dynamic CT
  Interventions: Procedure: Primovist-enhanced MRI

INTERVENTIONS:
Procedure: Primovist-enhanced MRI — Performance of Primovist-enhanced MRI in HCC patients with very early or early stage disease, but with no suspicious intrahepatic HCC lesions by liver dynamic CT.
  Other Names: Gadoxetic acid (Gd-EOB-DTPA, Primovist)-enhancecd MRI

SUMMARY:
Gadoxetic acid (Gd-EOB-DTPA, Primovist)-enhanced MRI can affect on BCLC staging during the initial staging workups of definite HCC patients with very early or early stage disease, but with no suspicious intrahepatic HCC lesions by liver dynamic CT.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the leading causes of cancer related death worldwide, and its incidence continues to rise even in the Europe and the United States. Recent advancements in early diagnosis and treatment modalities have significantly improved survival in HCC patients, but, only a small portion of them can receive curative treatments. Treatment decision making in HCC is guided by tumor stage, which can be also affected by tumor status at presentation.Thus, intrahepatic tumor status can be pivotal for treatment decision making and for determining prognosis in HCC patients, especially in possible candidates for curative treatment.

The current AASLD guideline recommends that HCC patients with typical HCC ≥1 cm by liver dynamic computed tomography (CT) do not require further investigation to confirm the presence of HCC, and that appropriate treatment can be initiated based on tumor stage. However, other intrahepatic HCC lesion which is not detected by liver dynamic CT can be additionally detected only by Primovist-enhanced MRI.Although few studies have evaluated the usefulness of Primovist-enhanced MRI in HCC patients,most of these studies have been limited by the lack of an evaluation of shift in HCC stage and by the inclusion of patients with suspicious intrahepatic HCC lesions that had been already detected by liver dynamic CT. Furthermore, given the poor prognosis of HCC patients with recurrence after curative treatments such as liver transplantation, surgical resection, or radiofrequency ablation (RFA),accurate staging workup is essential for intrahepatic HCC, especially in patients with a very early or early Barcelona Clinic Liver Cancer (BCLC) staged HCC. To date, however, no evidence based recommendations have been made regarding the benefit of add-on examination of Primovist-enhanced MRI during initial staging workups in HCC patients who are candidates for curative treatment after diagnosis by liver dynamic CT.

In this prospective multicenter study, therefore, we will assess the usefulness of Primovist-enhanced MRI during the initial staging workups of HCC patients with very early or early stage disease, but with no suspicious intrahepatic HCC lesions by liver dynamic CT. We will examine whether Primovist-enhanced MRI could provide additional information on BCLC stage, by directly comparing to liver dynamic CT in these patients. Furthermore, we assess whether add-on Primovist-enhanced MRI after a diagnosis of HCC by liver dynamic CT could aid treatment decision making in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age
* Patients who are initially diagnosed as having hepatocellular carcinoma with very early or early BCLC stage by liver dynamic CT at each hospital
* Performance status 0 or 1
* Child-Turcotte-Pugh score ≤8

Exclusion Criteria:

* Age of younger than 18
* Patients with any concurrent cancer other than hepatocellular carcinoma. Any cancer curatively treated at least 3 years prior to entry is permitted.
* Patients with BCLC B, C, or D staged HCC at initial diagnosis by liver dynamic CT
* Patients with suspicious intrahepatic malignant lesion by liver dynamic CT
* Patients with HIV infection
* Female patients in pregnancy
* Clinically hemodyanmically unstable patients
* Patients with previous life-threatening anaphylactic reaction to contrast media
* Patients scheduled for biopsy or liver surgery within 24 h post-administration of the study
* Patients who cannot underwent CT due to renal insufficiency (estimated GFR < 30 mL/min/1.73m2)
* Patients who cannot perform MRI due to contraindication of MRI (e.g. an implanted cardiac pacemaker)
* Patients in whom MRI was performed before liver dynamic CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients with very early (BCCLC stage 0) or early (BCLC stage A) stage disease, but with no suspicious intrahepatic HCC lesions by liver dynamic CT
Sampling Method: Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
incidence of change of BCLC stage after add-on Primovist-enhanced MRI in HCC patients with very early or early stage disease, but with no suspicious intrahepatic HCC lesions by liver dynamic CT. | Performance of Primovist enhanced MRI within the first 7 days after liver dynamic CT

SECONDARY OUTCOMES:
Incidence of newly detected intrahepatic HCC lesionss by Primovist-enhanced MRI, but, these lesions were not detected by liver dynamic CT | Performance of Primovist-enhacned MRI within 7 days after liver dynamic CT
Incidence of newly detected intrahepatic benign lesions by Primovist-enhanced MRI, but, these lesions were not detected by liver dynamic CT | Performance of Primovist-enhanced MRI within 7 days after liver dynamic CT
Frequency of change in treatment modality in patients with change of BCLC stage after Primovist-enhanced MRI | Performance of Primovist-enhanced MRI within 7 days after liver dynamic CT
Sensitivity, specificity, false positive predictive value, false negative predictive value, and accuracy of Primovist-enhanced MRI | after performance of Primovist-enhanced MRI and liver dynamic CT

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Woo Lee, M.D., Principal Investigator — Department of Internal Medicine, Inha University Hospital, Inha University School of Medicine, Incheon, Repubulic of Korea
Locations (1):
- Jin-Woo Lee, Incheon, South Korea